CLINICAL TRIAL: NCT03321552
Title: Percutaneous Deep Vein Arterialization Post-Market Study
Brief Title: PROMISE International
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LimFlow SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU PMS Revision 4.1
Record Dates: First submitted 2017-08-30; First posted 2017-10-25 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Critical Limb Ischemia
Keywords: Desert foot; No-option patients; Venous arterialization
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Percutaneous deep vein arterialization (Experimental): Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach
  Interventions: Procedure: Percutaneous deep vein arterialization; Device: LimFlow System

INTERVENTIONS:
Procedure: Percutaneous deep vein arterialization — Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach
Device: LimFlow System — Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach

SUMMARY:
The objective of this post-market study is to evaluate the safety and effectiveness of the LimFlow System in creating a below-the-knee arterio-venous fistula for venous arterialization in subjects with critical limb ischemia.

DETAILED DESCRIPTION:
This study will investigate the safety and effectiveness of the LimFlow System for creating an arterio-venous fistula in the below-the-knee vascular system using an endovascular, minimally invasive approach for the treatment of critical limb ischemia in subjects ineligible for conventional endovascular or surgical limb salvage procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 21 and < 95 years of age
* Clinical diagnosis of symptomatic critical limb ischemia, defined as Rutherford category 5 or 6
* Assessment that no conventional surgical or endovascular treatment is possible
* Proximally, the target in-flow artery at the cross-over point must be treatable with a 3.5 - 4.0 mm stent after pre-treatment (by visual estimate), and be <50% stenosed
* Subject is willing and has adequate support to comply with protocol requirements, including medication regimen and follow-up visits

Exclusion Criteria:

* Concomitant hepatic insufficiency, deep venous thrombus in target limb, uncorrected coagulation disorders, or current immunodeficiency disorder
* Prior vein stripping surgery and/or vessel harvesting for CABG in the limb intended for study
* Life expectancy less than 12 months
* Patient currently taking coumarin/warfarin which, in the opinion of the attending physician, interferes with the patient's treatment
* Any significant medical condition which, in the attending physician's opinion, may interfere with the patient's optimal treatment
* Patient currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this treatment
* Patient unable to give consent
* Pregnant or breastfeeding women
* Documented myocardial infarction or stroke within previous 90 days
* Patients suffering from renal insufficiency (GFR value less than 30 ml/min/1.73 m²) who are not on hemodialysis
* Patients with vasculitis and/or untreated popliteal aneurysms
* Patients with acute limb ischemia
* Prior peripheral arterial bypass procedure above or below the knee which could inhibit proximal inflow to the stent graft
* Lower extremity venous disease with significant edema in the target limb that may inhibit the procedure and/or jeopardize wound healing, in the investigator's opinion
* Known or suspected systemic or severe infection (e.g., WIfI foot Infection grade of 3)
* Known or suspected allergies or contraindications to stainless steel, nickel, or contrast agent that cannot be adequately pre-treated, or patients who cannot receive anticoagulation or antiplatelet aggregation therapy
* Severe heart failure, which in the opinion of the investigator may compromise subject's ability to safely undergo a percutaneous procedure (e.g., known ejection fraction of < 40%, NYHA Classification III-IV)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Universitätsklinikum Graz, Graz, Austria
- Germany (5):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad, Baden-Wurttemberg
  - Klinikum Arnsberg GmbH, Arnsberg, North Rhine-Westphalia
  - St. Franziskus-Hospital GmbH, Münster, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - St. Antonius Hospital, Nieuwegein
- Auckland City Hospital, Auckland, New Zealand
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Schreve MA, Lichtenberg M, Unlu C, Branzan D, Schmidt A, van den Heuvel DAF, Blessing E, Brodmann M, Cabane V, Lin WTQ, Kum S. PROMISE international; a clinical post marketing trial investigating the percutaneous deep vein arterialization (LimFlow) in the treatment of no-option chronic limb ischemia patient. CVIR Endovasc. 2019 Jul 31;2(1):26. doi: 10.1186/s42155-019-0067-z. PMID 32026120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 60 subjects screened at 10 sites in 4 countries resulting in 34 subjects enrolled between December 2017 and January 2022.
Pre-assignment Details: Subjects were screened by site personnel and once it was deemed they met inclusion and exclusion criteria, consent was obtained and imaging of the target arterial and venous anatomy were uploaded for review by an independent review committee to confirm that the patients were "no-option", i.e., with no capacity for standard endovascular or surgical treatment.
Period: Overall Study
Arm/Group | Percutaneous Deep Vein Arterialization
Started | 34 (There were 34 subjects enrolled with 35 legs treated.)
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 35 legs treated in 34 subjects enrolled
Units Other Than Participants: Legs
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
Number analyzed (Legs) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1
  Netherlands | 9
  Singapore | 4
  Germany | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Population: Collected for 32 subjects only
  kg/m²
    number analyzed (Participants) | 32
    (all) | 25.0 (4.4)
Current or former smoker [Count of Participants; unit: Participants] — Population: Smoking history unknown in 6 subjects
  Participants
    number analyzed (Participants) | 28
    (all) | 16
Diabetes [Count of Participants; unit: Participants] | 22
Hypertension requiring medication [Count of Participants; unit: Participants] — Population: Medical history characteristic unknown for 1 subject
  Participants
    number analyzed (Participants) | 33
    (all) | 26
Hyperlipidaemia requiring medication [Count of Participants; unit: Participants] — Population: Medical history characteristic unknown for 1 subject
  Participants
    number analyzed (Participants) | 33
    (all) | 23
Renal insufficiency [Count of Participants; unit: Participants]
  Any renal insufficiency | 11
  Renal insufficiency requiring dialysis | 6
Heart failure [Count of Participants; unit: Participants] | 18
Prior Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 10
Prior stroke [Count of Participants; unit: Participants] | 6
Prior intervention to target limb [Count of Units; unit: Legs] | 31
Rutherford classification [Count of Units; unit: Legs] — Rutherford's chronic limb ischemia classification consists of seven (7) categories:
  * 0 Asymptomatic
  * 1 Mild claudication
  * 2 Moderate claudication
  * 3 Severe claudication
  * 4 Ischemic rest pain
  * 5 Minor tissue loss
  * 6 Major tissue loss
  Legs
    Rutherford Class 5 | 31
    Rutherford Class 6 | 4

OUTCOME MEASURES:

1. Primary Outcome: Amputation-free Survival
Description: Freedom from death or major amputation as calculated using the Kaplan-Meier estimate
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
percentage of participants | 50.7 [32.5 to 66.3]

2. Secondary Outcome: Wound Healing
Description: Complete index wound healing as assessed by wound pictures
Time Frame: Throughout one year
Measure: Count of Units; unit: Legs
Units Other Than Participants: Legs
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 13
Number analyzed (Legs) | 14
Legs | 10

3. Secondary Outcome: Primary and Secondary Patency as Assessed by Duplex Ultrasound
Description: Stent graft patency as assessed by duplex ultrasound and calculated using the Kaplan-Meier estimate
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of legs
Units Other Than Participants: Legs
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 32
Number analyzed (Legs) | 33
percentage of legs
  Primary patency | 34.0 [14.6 to 54.5]
  Secondary patency | 67.4 [42.3 to 83.4]

4. Secondary Outcome: Limb Salvage
Description: Freedom from major amputation as calculated using the Kaplan-Meier estimate
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of legs
Units Other Than Participants: Legs
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
Number analyzed (Legs) | 35
percentage of legs | 66.6 [46.7 to 80.6]

5. Secondary Outcome: Deterioration in Renal Function
Description: Number of participants with deterioration in renal functionas assessed by changes in creatinine level
Time Frame: One month and six months
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
Participants
  Deterioration in renal function at 1 month | 0
  Deterioration in renal function at 2 months | 2

6. Secondary Outcome: Interventions With Technical Success (Procedure Completion)
Description: Procedure completion and immediate morphological success with successful placement of the arterial and venous catheters in the desired location in the limb, and ability to place the stent graft
Time Frame: Immediately post-procedure
Measure: Count of Units; unit: Interventions
Units Other Than Participants: Interventions
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
Number analyzed (Interventions) | 35
Interventions | 33

7. Secondary Outcome: Interventions With Procedural Success (Technical Success Without Death, Major Amputation, or Re-intervention)
Description: Combination of technical success without death, major amputation, or re-intervention
Time Frame: One month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 34
Participants | 24

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Percutaneous Deep Vein Arterialization
All-Cause Mortality (participants affected / at risk) | 7/34
Serious Adverse Events (participants affected / at risk) | 32/34
Other Adverse Events (participants affected / at risk) | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Deep Vein Arterialization (N=34)
Arterial or venous occlusion (target limb) (Vascular disorders) | 19 (28)
Wound infection (Infections and infestations) | 10 (14)
Pain (target limb) (Vascular disorders) | 7 (9)
Wound healing disorder (Vascular disorders) | 5 (6)
Myocardial infarction (Vascular disorders) | 4 (4)
Gangrene or necrosis (Vascular disorders) | 3 (3)
Sepsis or systemic infection (Infections and infestations) | 3 (3)
Cardiac rhythm disorder (Cardiac disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Stroke (Vascular disorders) | 2 (2)
Chest infection (Infections and infestations) | 1 (2)
Access site bleeding or hematoma (Surgical and medical procedures) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hypoglycemia or hyperglycemia (Endocrine disorders) | 1 (1)
New wound or ulcer (Vascular disorders) | 1 (1)
Pain (non-target limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute liver failure (Hepatobiliary disorders) | 1 (1)
Bowel ischemia (Vascular disorders) | 1 (1)
Erythema and tenderness (Vascular disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Deep Vein Arterialization (N=34)
Arterial or venous occlusion (target limb) (Vascular disorders) | 3 (3)
Pain (target limb) (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
PROMISE International was a post-market study of a CE-marked device and consisted of a single study arm due to the extreme nature of the alternative (i.e., major amputation). As such, all data reported are descriptive and are not statistically tested against any comparator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03321552/Prot_SAP_000.pdf